CLINICAL TRIAL: NCT03755401
Title: A Pilot Randomized Controlled Trial of Trauma-Focused Psychodynamic Psychotherapy (TFPP) at the VA in Veterans With PTSD
Brief Title: Post-Traumatic Stress Disorder Focused Psychodynamic Psychotherapy
Acronym: RCT of TFPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: VA New York Harbor Healthcare System (U.S. Federal Agency); Weill Medical College Clinical Science Translation Center (Unknown); American Psychoanalytic Association (APsA) (Unknown); International Psychoanalytic Association (IPA) (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-13720; 1UL1TR002384-02 (NIH); 1UL1TR002384 (NIH)
Record Dates: First submitted 2018-11-13; First posted 2018-11-28 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: PTSD
Keywords: psychotherapy; psychodynamic psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2,2,3,3-tetrafluoroputrescine; Psychotherapy, Psychodynamic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of psychosocial interventions
Who Masked: Outcomes Assessor
Masking Description: All assessments will be performed by blinded clinical assessors; randomization accomplished by computer algorhythm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TFPP (Experimental): TFPP is a manualized 16-24 session psychodynamic psychotherapy targeted on trauma symptoms of PTSD
  Interventions: Other: TFPP
- TAU (Active Comparator): TAU in this study is treatment for PTSD as currently delivered at the VA
  Interventions: Other: TAU

INTERVENTIONS:
Other: TFPP — Trauma-Focused Psychodynamic Psychotherapy
  Other Names: psychodynamic psychotherapy
  Arms: TFPP
Other: TAU — treatment as usual at the VA for PTSD
  Arms: TAU

SUMMARY:
This is a randomized controlled trial of Trauma-Focused Psychodynamic Psychotherapy (TFPP) in comparison with TAU (at the VA) in a 2:1 ratio in 75 Veterans with PTSD who have not responded to standard treatment at the VA.

DETAILED DESCRIPTION:
Veterans with PTSD are a highly vulnerable population with tremendous disability and unmet needs. Few VA patients with PTSD now actually receive evidence-based psychotherapy because current exposure-based treatments have low uptake. The project goal is to expand the range of PTSD psychotherapy treatments available at Veterans Administration Medical Centers. This pilot trauma recovery proposal takes the next step in translating a brief efficacious psychotherapy developed and tested for panic disorder, Panic Focused Psychodynamic Psychotherapy (PFPP) for Veterans with PTSD at the VA New York Harbor Healthcare System (VA NYHHCS). PFPP was developed, manualized, and studied in RCTs over the past two decades. We hope that Trauma-Focused Psychodynamic Psychotherapy (TFPP), an adaptation of PFPP, with its high response rates in panic disorder with/without agoraphobia, and non-exposure protocol, will fill crucial gaps in Veteran care. A major challenge facing psychotherapy research is translating and implementing efficacious therapies to the community. No psychodynamic psychotherapy for anxiety or PTSD has achieved this in the US. This pilot RCT represents a paradigm shift in its approach to trauma. TFPP will be the only PTSD treatment for Veterans to incorporate Veterans' input into refinement of the treatment as this project progresses. TFPP targets aspects of traumatic experience and approaches Veterans' lives more broadly than the symptom-focused treatments the VA currently offers our traumatized Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Reporting moderate PTSD, as defined by a CAPS score of >40
* Have at least one of the following history with CPT and/or PE:

  * offered and declined
  * dropped out of treatment
  * been determined unsuitable by their treatment team
  * received treatment but continue to experience symptoms meeting entrance criteria.
* Require stabilization on psychiatric medication for 2 month period prior to entry into study to avoid confounding treatments

Exclusion Criteria:

* Presence of SCID-5 assessed psychotic disorder, bipolar disorder, or substance use that would interfere with trial demands
* Severe suicidality that would require immediate crisis management
* Organic mental syndromes, delirium, or unstable medical conditions that would interfere with trial demands
* Inability to meet trial demands.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-11-02 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms as per DSM-5 as measured by CAPS-5 | baseline, 16 weeks (termination), 3 month follow-up
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). Low score indicates fewer PTSD symptoms, high score indicates more PTSD symptoms.

SECONDARY OUTCOMES:
Change in anxiety symptoms as measured by HARS. | baseline, 16 weeks (termination), 3 month follow-up
  Hamilton Anxiety Rating Scale (HARS). Low score indicates fewer state anxiety symptoms, high score indicates greater state anxiety symptoms
Change in reflective capacity as measured by RF score. | baseline, 16 weeks (termination), 3 month follow-up
  Reflective Function Scale (RF). Low score indicates poor ability to reflect on relationships and self, high score, indicates better capacity to reflect on others and self.
Change in depression symptoms as measured by HDRS. | baseline, 16 weeks (termination), 3 month follow-up
  Hamilton Depression Rating Scale (HDRS). Low score indicates few depressive symptoms, high score indicates high level of depressive burden (depression)
Change in mental and physical symptoms as measured by VR-12. | baseline, 16 weeks (termination), 3 month follow-up
  Veterans RAND 12-Item Health Survey (VR-12). The results of the VR-12 are summarized as two scores - a Mental Component Score (MCS) and a Physical Component Score (PCS). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS and MCS are both 50 points. The United States population standard deviation is 10 points. Therefore, each increment of 10 points above or below 50 corresponds to one standard deviation away from the population average.
Change in work and social adjustment as measured by WSAS. | baseline, 16 weeks (termination), 3 month follow-up
  Work and Social Adjustment Scale (WSAS). Low score indicates good social and work adjustment, high score indicates impairment socially and at work.
Change in degree of limitation in ability to work as measured by WLQ | baseline, 16 weeks (termination), 3 month follow-up
  Work Limitations Questionnaire (WLQ). Low score indicates few limitations at work, high score indicates many limitations at work
Childhood abuse history and trauma with CTQ | baseline
  Childhood Trauma Questionnaire (CTQ). Several different domains: Emotional Abuse: None=5-8; Low=9-12; Moderate=13-15; Severe=16+ Physical Abuse: None=5-7; Low=8-9; Moderate=10-12; Severe=13+ Sexual Abuse: None=5; Low=6-7; Moderate=8-12; Severe=13+ Emotional Neglect: None=5-9; Low=10-14; Moderate=15-17; Severe=18+ Physical Neglect: None=5-7; Low=8-9; Moderate=10-12; Severe=13+
Change in adult separation anxiety symptoms as measured by the SCI-SAS | baseline, 16 weeks (termination), 3 month follow-up
  Separation anxiety-child and adult measure rating scale (SCI-SAS). Separate scores generated for childhood separation anxiety and adult separation anxiety. Low scores indicate few separation anxiety symptoms, high scores indicate large separation anxiety burden.
Assessment of life events on LEC. | baseline
  Life Events Checklist (LEC). No composite score-tracks traumatic life events

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Milrod, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- VA New York Harbor Healthcare System - Manhattan Campus, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Busch FN, Milrod BL. Trauma-Focused Psychodynamic Psychotherapy. Psychiatr Clin North Am. 2018 Jun;41(2):277-287. doi: 10.1016/j.psc.2018.01.005. PMID 29739526
- [Result] Kehn M, Milrod B, Chen CK. Clinical Case of Trauma-Focused Psychodynamic Psychotherapy for a Veteran With PTSD and Race-Based Trauma. Am J Psychother. 2024 Sep 1;77(3):146-150. doi: 10.1176/appi.psychotherapy.20230040. No abstract available. PMID 39277802